CLINICAL TRIAL: NCT07062588
Title: A Phase 2, Multi-center, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study to Evaluate the Safety and Efficacy of AGA2115 in Adults With Type I, III, or IV Osteogenesis Imperfecta (OI)
Brief Title: Osteogenesis Imperfecta Trial of AGA2115 for ADUlts With COL1A1 and/or COL1A2 GeNetic Variations (IDUN)
Acronym: IDUN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Angitia Incorporated Limited (Industry)
Responsible Party: Sponsor
Organization: Angitia Biopharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT24-001
Record Dates: First submitted 2025-07-01; First posted 2025-07-14 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Osteogenesis Imperfecta (OI)
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AGA2115 Dose Regimen 1 (Experimental): Participants that complete the double-blind period receiving AGA2115 Dose 1 from study start to Month 12 will continue to a 12-month open-label period. Participants will then receive AGA2115 Dose 2 for Months 12 to 24.
  Interventions: Drug: AGA2115
- AGA2115 Dose Regimen 2 (Experimental): Participants that complete the double-blind period receiving AGA2115 Dose 2 from study start to Month 12 will continue to a 12-month open-label period. Participants will be kept on the same AGA2115 dose for Months 12 to 24.
  Interventions: Drug: AGA2115
- AGA2115 Dose Regimen 3 (Experimental): Participants that complete the double-blind period receiving AGA2115 Dose 3 from study start to Month 12 will continue to a 12-month open-label period. Participants will receive the same AGA2115 dose for Months 12 to 24.
  Interventions: Drug: AGA2115
- Placebo (Placebo Comparator): Participants that complete the double-blind period receiving placebo from study start to Month 12 will continue to a 12-month open-label period. Participants will receive AGA2115 Dose 3 for Months 12 to 24.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AGA2115 — Subcutaneous injection
  Arms: AGA2115 Dose Regimen 1; AGA2115 Dose Regimen 2; AGA2115 Dose Regimen 3
Other: Placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
This study will determine the effect of treatment of AGA2115 in adults with Type I, III, or IV osteogenesis imperfecta versus placebo.

DETAILED DESCRIPTION:
This Phase 2 dose-ranging study will evaluate the safety and efficacy of AGA2115 at a range of doses in adults with Type I, III, or IV osteogenesis imperfecta. The study will last 27 months with a 24-month treatment period and a 3-month follow-up period. During the first 12 months of the study, participants will be randomized 1:1:1:1 to receive either placebo or one of three dose levels of AGA2115 doses; treatment assignment will be double-blind. Months 12 to 24 will be open-label, and all participants will receive AGA2115. Participants will attend visits where safety and efficacy parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults (aged 18 to 75 years inclusive) with a clinical diagnosis of osteogenesis imperfecta Type I, III, or IV with documented genetic testing confirmation of genetic variations in the COL1A1 or COL1A2 genes
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol
* BMD T-score of ≤ -1.0 at the lumbar spine, total hip, or femoral neck

Exclusion Criteria:

* Vitamin D deficiency
* Concomitant uncontrolled diseases or conditions that could affect bone metabolism such as hypo-/hyperparathyroidism, hypo-/hyperthyroidism, abnormal thyroid function or thyroid disease, or other endocrine disorders
* Current hyper- or hypocalcemia
* History of rickets or osteomalacia or any skeletal condition (other than OI) leading to long-bone deformities and/or increased risk of fractures
* Treatment with bisphosphonates within the past 6 months
* Treatment with teriparatide, abaloparatide, strontium ranelate, or hormone replacement therapy within the past 12 months
* Treatment with denosumab (or denosumab biosimilars) within the past 2 years
* Treatment with anti-sclerostin antibody medications (romosozumab, setrusumab, blosozumab) at any time
* History of myocardial infarction or stroke (or other cardiovascular associated event deemed significant) within the past 12 months
* Malignancy within the last 5 years
* Pregnant or breastfeeding women, or women planning to become pregnant during the study
* Participation in any clinical study within the past 12 months during which the participant was administered any IP (participant must also agree not to enroll in any other clinical study concurrently in which IP is administered)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Percent change from Baseline at Month 12 in lumbar spine BMD | 12 months

SECONDARY OUTCOMES:
Percent change from Baseline at Month 3 and 6 in lumbar spine, total hip, femoral neck, one-third distal radius, and total body (minus head) BMD | 3 and 6 months
Percent change from Baseline at Month 12 in total hip, femoral neck, one-third distal radius, and total body (minus head) BMD | 12 months
Percent change from Baseline at Week 1 and Month 1, 3, 6, 9, and 12 in P1NP and CTX-1 | Week 1, Month 1, 3, 6, 9, and 12
Percentage of participants with fractures during the double-blind treatment period | up to 12 months
Annualized fracture rate for incident fractures occurring during the double-blind treatment period (total, long-bone, vertebral, peripheral) | up to 12 months

OTHER OUTCOMES:
Assessment of TEAEs (collection and documentation of all adverse events occurring during the study) | Baseline to 24 months
Evaluation of AGA2115 observed serum concentration levels for the AGA2115 treatment groups | Baseline to 24 months
Number of participants who develop anti-AGA2115 antibodies | Baseline to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ann Zovein, MD, Study Director — Angitia Incorporated Limited
Locations (26):
- United States (10):
  - Phoenix Children's, Phoenix, Arizona
  - Yale University School of Medicine, New Haven, Connecticut
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Indiana University School of Medicine, Department of Medicine and Pediatrics Division of Endocrinology, Indianapolis, Indiana
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - University of Nebraska Medical Center (UNMC) - Diabetes and Endocrinology Center, Omaha, Nebraska
  - New Mexico Clinical Research & Osteoporosis Center, Inc. (NMCROC), Albuquerque, New Mexico
  - The Ohio State University Wexner Medical Center (OSUWMC), Columbus, Ohio
  - Oregon Health & Science University (OHSU) - The Harold Schnitzer Diabetes Health Center (HSDHC) - Endocrinology Clinic, Portland, Oregon
  - Vanderbilt University Medical Center (VUMC) - Eskind Diabetes Clinic, Nashville, Tennessee
- Instituto de Investigaciones Metabolicas Dr. Zanchetta - Sede Centro, Buenos Aires, Argentina
- Australia (4):
  - Monash University-Monash Medical Centre (MMC), Melbourne
  - Royal Melbourne Hospital, Parkville
  - Royal North Shore Hospital (RNSH), Saint Leonards
  - Adults Westmead Hospital, Westmead
- University Health Network - Toronto General Hospital - Osteoporosis Clinic, Toronto, Ontario, Canada
- Denmark (2):
  - Aarhus Universitetshospital - Medicinsk Endokrinologisk Afdeling (MEA) Ambulatoriet - Tage-Hansens Gade, Aarhus
  - Odense Universitetshospital, Odense
- France (2):
  - Hopital Edouard Herriot, Lyon
  - Assistance Publique-Hopitaux de Paris (AP-HP) - Hopital Lariboisiere, Paris
- Netherlands (3):
  - Leiden University Medical Center (LUMC) - Centrum voor botkwaliteit, Leiden
  - Erasmus MC, Rotterdam
  - Isala ziekenhuizen, Zwolle
- United Kingdom (3):
  - Cambridge University Hospitals NHS Foundation Trust-Addenbrooke's Hospital, Cambridge
  - Lothian Health Board, Western General Hospital, Edinburgh
  - Royal National Orthopaedic Hospital NHS Trust, London